CLINICAL TRIAL: NCT06291779
Title: Development of Pancreatic Cancer Diagnostic Method by Using a Reagent for Analyzing Purine Metabolite (Hypoxanthine, Xanthine) in Urine
Brief Title: Diagnosis of Pancreatic Cancer by Purine Metabolite (Hypoxanthine, Xanthine) in Urine
Status: Recruiting | Type: Observational
Sponsor: Ho-Seong Han (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor-Investigator, Ho-Seong Han, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: SNUBH-GS- HBP5; E-2211-792-350 (local IRB) (Other: Seoul National University Bundang Hospital)
Record Dates: First submitted 2023-01-14; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Pancreas Cancer; Diagnosis
Keywords: Pancreatic cancer; hypoxanthine/xanthine concentration in urine
MeSH Terms: conditions — Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — measurement of hypoxanthine and xanthine concentrations in urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic cancer group: scheduled for curative surgery for pancreatic cancer
  Interventions: Device: Purine metabolite (Hypoxanthine, Xanthine) in urine by CubeBio
- Control group: group included healthy individuals as well as patients with benign diseases
  Interventions: Device: Purine metabolite (Hypoxanthine, Xanthine) in urine by CubeBio

INTERVENTIONS:
Device: Purine metabolite (Hypoxanthine, Xanthine) in urine by CubeBio — * Collect urine from the patient to measure urinary hypoxia, xanthine concentration.
  * Hypoxic acid, xanthine analysis in urine using High Performance Liquid Chromatography (HPLC).
  * After that, hypoxanthine and xanthine will be analyzed using purine metabolite analysis reagents.
  * Compare the cutoff of the metabolic value of Pancreas cancer clarified in the existing research and the value of the sample.

SUMMARY:
* This study aim to develope a diagnostic method of pancreatic cancer by using a reagent for analyzing purine metabolite (Hypoxanthine, Xanthine) in urine.
* It is safe and cost effective compare to radiologic or blood test. It can be used for initial screening test for healty population.

DETAILED DESCRIPTION:
* CubeBio and Seoul National University Bundang Hospital signed a joint technology development agreement to compare the analytical performance of existing analytical methods and purine metabolite analysis reagents developed by CubeBio.
* Through quantitative analysis of hypoxanthine and xanthine in the urine of normal people and pancreatic cancer patients, we plan to confirm the possibility of diagnosing pancreatic cancer using reagents for analyzing purine metabolites.
* Early diagnosis of pancreatic cancer is a key determinant of cure and survival rates, and impact on all aspects of cancer, including rate of progression, treatment, and prognosis.
* This study could change the paradigm of pancreatic cancer screening by evaluating the stability and accuracy of urinary purine metabolite analysis reagents.

ELIGIBILITY:
1. pancreatic cancer group

   Inclusion Criteria:
   * Pancreatic ductal adenocarcinoma that is pathologically confirmed or shows characteristic radiologic features
   * Patients with resectable pancreatic cancer at the time of surgery (Including borderline resectable pancreatic cancer at the time of diagnosis or Locally advanced pancreatic cancer after chemotherapy or radiation therapy)
   * Patients without invasion of adjacent organs other than the left adrenal gland and mesocolon
   * Patients with informed consent

   Exclusion Criteria:
   * History of other malignancy (Inclusive if there is no evidence of recurrence after 5 years of treatment)
   * Patient with Inflammatory disease(e.g. severe pancreatitis, cholangitis)
   * Patients with underlying diseases at high risk of general anesthesia
   * Other subject whom the investigator deems inappropriate
2. control group Inclusion Criteria included healthy individuals as well as patients with benign diseases.

Exclusion criteria for the control group included a previous cancer diagnosis within the past five years, active inflammatory diseases, borderline malignant pancreatic tumors, or a postoperative pathological finding of malignancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer group: comprised patients who were scheduled for curative surgery for pancreatic cancer
  Control group: The control group included healthy individuals as well as patients with benign diseases
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-02-26 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Urine | 1 day
  mean concentration of purine metabolites in urine

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Seong Han, M.D. Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Ho-Seong Han, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Wu H, Xue R, Dong L, Liu T, Deng C, Zeng H, Shen X. Metabolomic profiling of human urine in hepatocellular carcinoma patients using gas chromatography/mass spectrometry. Anal Chim Acta. 2009 Aug 19;648(1):98-104. doi: 10.1016/j.aca.2009.06.033. Epub 2009 Jun 21. PMID 19616694